CLINICAL TRIAL: NCT00858975
Title: Study of Cryotherapy for Renal Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yeong-Shiau Pu, Department of Urology / National Taiwan University Hospital
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200709063R
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2012-12

CONDITIONS: Renal Tumors
Keywords: renal tumor; cryotherapy; cytokine
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryotherapy (Experimental): The patients who receive cryotherapy for their renal tumors
  Interventions: Procedure: cryotherapy

INTERVENTIONS:
Procedure: cryotherapy — Placing 4-6 cryotherapy probes into the renal tumors and conducting two cycles of freezing and thawing

SUMMARY:
The purpose of this study is to study the change of tumor size and serum cytokine in the patients who received cryotherapy for the renal tumors.

ELIGIBILITY:
Inclusion Criteria:

* The patients who have renal tumor less than 7 cm and receive cryotherapy

Exclusion Criteria:

* The tumor size is larger than 7 cm
* The patients do not approve the surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Tumor size | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan